CLINICAL TRIAL: NCT05320783
Title: Effect on Music Therapy on Quality of Recovery and Postoperative Pain After Gynecological Laparoscopy
Brief Title: Effect on Music Therapy on Quality of Recovery After Gynecological Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eun Kyung Choi (Other)
Responsible Party: Sponsor-Investigator, Eun Kyung Choi, Professor, Yeungnam University College of Medicine
Organization: Yeungnam University College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YUMC 2019-09-052
Record Dates: First submitted 2022-03-15; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Quality of Recovery After General Anesthesia; Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music intervention (Active Comparator): Headphone was placed on the each patient. The classical music was started to the patients with individual comfortable volume.
  Interventions: Other: music
- control (Placebo Comparator): Headphone was placed on the each patients, but the music player was not started.
  Interventions: Other: control

INTERVENTIONS:
Other: music — Classical music pre-selected was started to the patients with individual comfortable volume.
  Arms: music intervention
Other: control — music player was not started.
  Arms: control

SUMMARY:
In the present study, we intended to evaluate the effect of music intervention on postoperative pain, nausea, and comprehensive recovery quality in patients undergoing gynecological laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status classification I and II,
* undergoing gynecological laparoscopic surgery

Exclusion Criteria:

* Any hearing impairment,
* Known psychiatric or memory disorder
* Alcohol or analgesics abuse
* Inability to complete quesationnaires

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Recovery quality | At postoperative day, 1
  Patient-reported survery, quality of recovery 40 (QoR 40): sum scores range from 40 to 200 (40; poor ~ 200; excellent quality of recovery)
Postoperative pain | 36 hours after surgery
  Numeric rating scale (NRS, 0-10)O; no pain ~ 10; the most severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Eun kyung Choi, Daegu, Korea (the Republic Of), South Korea

IPD SHARING:
Plan to Share IPD: Yes